CLINICAL TRIAL: NCT04696016
Title: Guiding Sufentanil Administration With Skin Conductance in Mechanically Ventilated Intensive Care Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P2020/402 / B4062020000124
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Nociceptive Pain
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin conductance guided (Experimental): Sufentanil is titrated by the intensive care team to maintain skin conductance in target
  Interventions: Procedure: Skin conductance guided antinociception
- Standard care (Active Comparator): Sufentanil is titrated at the discretion of the intensivist
  Interventions: Procedure: Standard care antinociception

INTERVENTIONS:
Procedure: Skin conductance guided antinociception — The value of skin conductance guides the titration of sufentanil
  Arms: Skin conductance guided
Procedure: Standard care antinociception — The intensive care team titrates antinociception based on their standard approach (using a clinical approach by assessing blood pressure, heart rate, and ventilator dyssynchrony).
  Arms: Standard care

SUMMARY:
Opioid administration in mechanically ventilated patients in the intensive care unit (ICU) is essential to maintaining patient respiratory and hemodynamic stability. Mechanical ventilation is a persistently nociceptive event that can continuously causes discomfort in the trachealy intubated patient. This can lead to patient-ventilator dyssynchrony, tachycardia, hypertension, and their associated complications. Opioids blunt respiratory drive, which facilitates mechanical ventilation, and decrease the sympathetic response to nociception. However, excessive opiate administration is associated with many adverse events, including respiratory depression, delirium, ileus, nausea, and vomiting. Currently, the standard administration in our institution of sufentanil, a potent opiate, consists of continuous infusions of 0.15µg/kg/h to 0.3µg/kg/h.

Mechanically ventilated patients are unable to speak and are often sedated. This greatly impacts the patient's capacity to communicate pain. The use of a nociceptive monitor may be a possible solution. Skin conductance monitoring (Pain Monitor, Med-Storm, Norway), measures the peaks per second of electrical conduction. This non hemodynamic monitor uses skin conduction as a surrogate to nociception (i.e., the patient's unconscious response to a noxious stimulus). It may consequently guide opioid administration in ICU patients towards and avoid the consequences of excessive or inadequate antinociception.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient admitted to the ICU requiring endotracheal intubation, antinociception, and sedation

Exclusion Criteria:

* Traumatic brain injury
* use of ketamine, dexmedetomidine, or clonidine
* pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of sufentanil requirements | one day to 2 weeks
  Sufentanil requirements (µg/kg/h)

SECONDARY OUTCOMES:
Concentration of propofol requirements | one day to 2 weeks
  Propofol requirements (mg/kg/h)
Concentration of noradrenaline requirements (concentration of) | one day to 2 weeks
  noradrenaline requirements (µg/kg/min)
Intubation time | one day to 2 weeks
  Total time of mechanical ventilation (intubated)
Composite post extubation related complications | one day to 2 weeks
  post extubation opioid related complications (e.g., delirium, vomiting, nausea, ileus, respiratory acidosis, hypoxemia, reintubation).

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Taccone, Principal Investigator — Université Libre de Bruxelles

IPD SHARING:
Plan to Share IPD: Undecided